CLINICAL TRIAL: NCT04155957
Title: Evaluation of Safety and Efficacy of ReHub in Patients Who Underwent Primary Total Knee Arthroplasty
Acronym: REHAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bio-Sensing Solutions S.L. (DyCare) (Industry)
Collaborators: Hospital Clinic of Barcelona (Other); EASME (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCEB28042019
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation Group (Active Comparator): Participants follow the usual fast-track protocol used at Hospital Clínic de Barcelona for Total Knee Arthroplasty and perform a daily 5-exercise plan autonomously.
  Interventions: Other: Rapid Recovery Rehabilitation Programme
- ReHub Group (Experimental): Participants follow the usual fast-track protocol used at Hospital Clínic de Barcelona for Total Knee Arthroplasty but use the telerehabilitation platform ReHub to do the exercises in their rehabilitation plan at home and to have their progress monitored.
  Interventions: Other: Rapid Recovery Rehabilitation Programme; Device: ReHub

INTERVENTIONS:
Other: Rapid Recovery Rehabilitation Programme — Usual intervention at Hospital Clínic de Barcelona for post-operative rehabilitation of TKA patients. Participants, already at home after hospital discharge, must perform 5 different exercises 4 times a day (twice in the morning, twice in the afternoon).
  Participants are also encouraged to walk and stretch their legs. Domiciliary visits by a physiotherapist start at approximately 2 weeks after the surgery to help participants do the exercises.
Device: ReHub — Participants use a telerehabilitation platform, ReHub, as a guide to perform the TKA rehabilitation exercises of the Rapid Recovery Rehabilitation Programme intervention.
  The exercise plan in ReHub is carried out by a site physiotherapist on the first day after discharge by using ReHub to acquire the participant's movement pattern with a wearable inertial sensor that transmits data to the platform.
  The wearable inertial sensor participants must wear tracks movement while they do the TKA rehabilitation exercises. Movement is analysed and feedback is given in real time. At the end of each exercise, participants can select if they have felt pain in a scale from 1 to 10. A physiotherapist monitors the participants' progress remotely.
  Arms: ReHub Group

SUMMARY:
This is a randomized, non-blinded, parallel assignment, clinical trial for the evaluation of safety and efficacy of ReHub, a telerehabilitation system made up of a cloud platform and an exercise kit with smart sensors, for performing rehabilitation exercises after a primary Total Knee Arthroplasty.

Primary TKA patients are allocated randomly to the control arm or the experimental arm with a 1:1 ratio. Both arms follow the usual rapid recovery protocol for TKA surgeries at Hospital Clínic de Barcelona, which includes discharge after 2-3 days from the surgery, the prescription of a daily plan of 5 exercises for autonomous rehabilitation and domiciliary visits by a physiotherapist starting approximately 2 weeks after the surgery. The experimental arm participants use ReHub to do their exercises instead of working independently and physiotherapists monitor their performance and adherence remotely.

Outcomes assessment is performed at hospital discharge (baseline), at stitch removal (2 weeks after baseline) and 2 weeks after stitch removal (4 weeks after baseline).

ELIGIBILITY:
Inclusion Criteria:

* Candidates to primary TKA
* Age from 18 to 75 years old
* Ability to understand and accept the clinical study procedure and to sign an informed consent form
* Good predisposition to the use of technology or cohabitation with someone that can give them technological support
* Availability to attend the Hospital for control visits
* Patient resides in the area of influence of Hospital Clínic de Barcelona

Exclusion Criteria:

* Reluctance or inability to use technology
* Any type of disability that could alter the homogeneity of the study
* Sensory and/or cognitive impairment
* Concomitant medical conditions that may influence the rehabilitation process
* Any local or systemic complications after TKA surgery (e.g. surgical wound infection, suspicious of deep vein thrombosis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Active Knee Range of Motion (º) | Baseline, 2 weeks and 4 weeks after discharge
  Range of motion of the replaced knee without the aid of the outcomes assessor will be measured with a conventional goniometer.

SECONDARY OUTCOMES:
Change in the Timed Up-and-Go test score (s) | Baseline, 2 weeks and 4 weeks after discharge
  The TUG test outcome is the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Change in Self-Reported Pain Level: Visual Analogue Scale | Baseline, 2 weeks and 4 weeks after discharge
  The pain level will be reported by the participant with a Visual Analogue Scale from 0 to 10, with 0 being the absence of pain and 10 being the worst pain imaginable.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Baseline, 2 weeks and 4 weeks after discharge
  Scores for the WOMAC questionnaire range from 0 to 96, with 0 being the best state and 96 the worst state.
Change in EuroQol-5D-5L (EQ-5D-5L) score | Baseline, 2 weeks and 4 weeks after discharge
  Scores for the EQ-5D-5L questionnaire are 5-digit numbers, each one representing a different aspect of quality of life. Digits can range from 1 to 5. 11111 is considered the ideal state and 55555 the worst state. 9 is used for absent or non-valid answers. The questionnaire also includes a Visual Analogue Scale for indicating perceived self's health state in a scale from 0 (worst state) to 100 (best state).
Change in Quadriceps Strength (kg) | Baseline, 2 weeks and 4 weeks after discharge
  Strength of the quadriceps in the intervened leg will be measured with a dynamometer.
Change in Hamstring Strength (kg) | Baseline, 2 weeks and 4 weeks after discharge
  Strength of the hamstring muscles in the intervened leg will be measured with a dynamometer.
Satisfaction with ReHub: System Usability Scale | 4 weeks after discharge
  Measured with the score from the System Usability Scale questionnaire, which can range from 0 (worst result) to 100 (best result). Only for participants in the experimental arm.
Change in Passive Knee Range of Motion (º) | Baseline, 2 weeks and 4 weeks after discharge
  Range of motion of the replaced knee with the aid of the outcomes assessor will be measured with a conventional goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Salvi Prat Fabregat, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Nuevo M, Mahdavi H, Rodriguez D, Faura T, Fabrellas N, Balocco S, Conti M, Castagna A, Prat S. Evaluation of Safety and Efficacy of ReHub in Patients Who Underwent Primary Total Knee Arthroplasty: Study Protocol for a Randomized Controlled Trial. Int J Surg Protoc. 2021 Apr 19;25(1):34-41. doi: 10.29337/ijsp.138. PMID 34013143